CLINICAL TRIAL: NCT06659757
Title: A Single-Centre, Double-Blinded, Randomised, Placebo-Controlled Phase I Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of KIT2014 in Healthy Subjects.
Brief Title: A Study to Investigate the Safety and Tolerability of Single and Multiple Ascending Doses of KIT2014 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kither Biotech Srl (Industry)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: KIT2014-01
Record Dates: First submitted 2024-10-22; First posted 2024-10-26 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A: Single Ascending Dose (SAD) (Experimental): Healthy volunteers - Up to 4 dose levels of KIT2014 will be evaluated in Part A. Dose levels will be investigated in sequential cohorts (A1 to A4) of 8 healthy participants per cohort (ratio 3:1 active:placebo).
  Interventions: Drug: KIT2014; Other: Placebo
- Part B: Multiple Ascending Dose (MAD) (Experimental): Healthy volunteers - Up to 3 dose levels of KIT2014 will be evaluated in Part B. Dose levels will be investigated in sequential cohorts (B1 to B3) of 8 healthy participants per cohort (ratio 3:1 active:placebo).
  Interventions: Drug: KIT2014; Other: Placebo

INTERVENTIONS:
Drug: KIT2014 — KIT2014 will be administered by inhalation with a nebuliser
Other: Placebo — Placebo will be administered by inhalation with a nebuliser

SUMMARY:
This is the first-in-human study with KIT2014 designed to provide safety, tolerability and pharmacokinetic data in healthy volunteers.

DETAILED DESCRIPTION:
This is a double-blind, randomised, placebo-controlled study to assess the safety, tolerability, and pharmacokinetics of ascending doses of inhaled KIT2014 administered via nebulizer to healthy adult participants. The study will be conducted in 2 parts, Part A (single ascending dose, SAD) and Part B (multiple ascending doses, MAD).

ELIGIBILITY:
Major Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are performed and must be able to understand the full nature and purpose of the study, including possible risks and adverse effects.
2. Adult males and females, 18 to 55 years of age (inclusive) at screening.
3. BMI ≥ 18.0 and ≤ 32.0 kg/m2, with a body weight of at least 60 kg for males and 50 kg for females.
4. Medically healthy, as determined by pre-study medical history, and without clinically significant abnormalities.
5. Normal spirometry results at Screening based on FEV1 ≥ 80% of predicted, FVC ≥ 80% of predicted and FEV1/FVC ratio ≥0.70.

Major Exclusion Criteria:

1. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic, psychiatric, or neurological disease/disorder, including any acute illness, determined by the PI to be clinically relevant.
2. Any respiratory infection or relevant respiratory problem within 14 days of Day 1.

Other inclusion/exclusion eligibility criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs), serious adverse events (SAEs) | Up to 10 days post-dose in SAD and up to 14 days after the last dose in MAD
  Incidence, type, severity, and relationship of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) after single and multiple inhaled administration of KIT2014 in healthy male and female participants.

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No